CLINICAL TRIAL: NCT01299571
Title: An Open Label, Multi-centre, Non-interventional Post-marketing Surveillance to Monitor the Safety and/or Efficacy of AVODART(Dutasteride) Administered in Korean BPH(Benign Prostatic Hyperplasia) Patients According to the Prescribing Information
Brief Title: AVODART(Dutasteride) Post-marketing Surveillance(PMS)
Acronym: AVO PMS
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 105194
Record Dates: First submitted 2011-02-17; First posted 2011-02-18 (Estimated); Results first posted 2011-04-18 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-06

CONDITIONS: Benign Prostatic Hyperplasia; Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Dutasteride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dutasteride: Patients administrated dutasteride at the site
  Interventions: Drug: Dutasteride

INTERVENTIONS:
Drug: Dutasteride — Basically there is no treatment allocation. Subjects who would be administered of dutasteride at their physicians' discretion will be enrolled. Dosage regimen will be recommended according to the prescribing information. Subjects will be enrolled consecutively.

SUMMARY:
An open label, multi-centre, non-interventional post-marketing surveillance to monitor the safety and/or efficacy of AVODART administered in Korean BPH patients according to the prescribing information

ELIGIBILITY:
Inclusion Criteria:

* The Korean BPH Patients administrated dutasteride according to the prescribing information

Exclusion Criteria:

* women and children and adolescents.
* patients with hypersensitivity to dutasteride, other 5-alpha reductase inhibitors, or any of the excipients.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The Korean BPH Patients administrated dutasteride
Sampling Method: Probability Sample
Enrollment: 3977 (Actual)
Dates: Start 2004-12; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The objective of this post-marketing surveillance (PMS) study was to assess the occurrence of adverse events reported after administration of Avodart in Korean benign prostatic hyperplasia (BPH) patients.
Groups:
- Avodart 0.5 mg: Avodart capsule containing 0.5 milligrams (mg) of dutasteride was administered orally once daily.
Period: Overall Study
Arm/Group | Avodart 0.5 mg
Started | 3977
Completed | 3870
Not Completed | 107
Not completed — Protocol Violation | 107

BASELINE CHARACTERISTICS:
Arm/Group | Avodart 0.5 mg
Number analyzed (Participants) | 3870
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline characteristics were collected in members of the Intent-to-Treat (ITT) Population, comprised of all participants who had been administered the investigational drug at least once and had completed safety assessments.
  Years | 67.3 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline characteristics were collected in members of the ITT Population, comprised of all participants who had been administered the investigational drug at least once and had completed safety assessments.
  Participants
    Female | 0
    Male | 3870
Race/Ethnicity, Customized [Number; unit: participants] — Baseline characteristics were collected in members of the ITT Population, comprised of all participants who had been administered the investigational drug at least once and had completed safety assessments.
  participants
    Korean | 3870
    Not Korean | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Adverse Event
Description: An adverse event is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. For a list of all adverse events occurring during the course of the study, see the table entitled "Other (Non-Serious) Adverse Events" in the Adverse Event section of the results record.
Time Frame: 6 months
Population: Intent-to-Treat (ITT) Population: all participants who had been administered the investigational drug at least once and had completed all safety assessments
Measure: Number; unit: participants
Groups:
- Avodart 0.5 mg: Avodart capsule containing 0.5 mg of dutasteride was administered orally once daily
Arm/Group | Avodart 0.5 mg
Number analyzed (Participants) | 3870
participants | 146
Statistical Analysis 1: Comparison: Avodart 0.5 mg; Test type: Superiority or Other; Percentage of participants = 3.8, 95% CI [3.2 to 4.4] — The estimated value represents the percentage of participants with adverse events

2. Secondary Outcome: Number of Participants With a Serious Adverse Event
Description: A serious adverse event is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or results in prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect. For a list of all serious adverse events occurring during the course of the study, see the table entitled "Serious Adverse Events" in the Adverse Event section of the results record.
Time Frame: 6 months
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Avodart 0.5 mg
Number analyzed (Participants) | 3870
participants | 5

3. Secondary Outcome: Number of Participants With the Indicated Unexpected Adverse Events
Description: An adverse event is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Unexpected adverse events include those not listed in the approved product information and not described as precautions or warnings.
Time Frame: 6 months
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Avodart 0.5 mg
Number analyzed (Participants) | 3870
participants
  Insomnia | 2
  Mouth Dry | 3
  Constipation | 2
  Abdominal Pain | 2
  Diarrhea | 2
  Vomiting | 1
  Colonic Polyp | 1
  Epigastric Discomfort | 1
  Gastroesophageal Reflux | 1
  Hemorrhoids | 1
  Asthenia | 1
  Fever | 1
  Chills | 1
  Pain | 1
  Spasms | 1
  Orofacial Dyskinesia | 1
  Embolism Pulmonary | 1
  Thrombosis Cerebral | 1
  Nose Congestion | 1
  Pneumonia | 1
  Lung Carcinoma | 1
  Skin Eruption | 1
  Thrombosis Venous Deep | 1

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events were coded by using World Health Organization Adverse Reactions Terminology (WHOART, preferred term level) according to the local regulation.
Arm/Group | Avodart 0.5 mg
Serious Adverse Events (participants affected / at risk) | 5/3870
Other Adverse Events (participants affected / at risk) | 146/3870
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avodart 0.5 mg (N=3870)
Diarrhea (Gastrointestinal disorders) | 1
Embolism Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1
Thrombosis Cerebral (Blood and lymphatic system disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Lung Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avodart 0.5 mg (N=3870)
Impotence (Psychiatric disorders) | 72
Libido Decreased (Psychiatric disorders) | 49
Ejaculation Disorder (Reproductive system and breast disorders) | 30
Dyspepsia (Gastrointestinal disorders) | 6
Gynaecomastia (Endocrine disorders) | 5
Mouth Dry (Gastrointestinal disorders) | 3
Insomnia (Psychiatric disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Colonic Polyp (Gastrointestinal disorders) | 1
Epigastric Discomfort (Gastrointestinal disorders) | 1
Gastroesophageal Reflux (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Localized Edema (General disorders) | 1
Asthenia (General disorders) | 1
Allergy (General disorders) | 1
Fever (General disorders) | 1
Chills (General disorders) | 1
Pain (General disorders) | 1
Dizziness (Nervous system disorders) | 2
Spasms (Nervous system disorders) | 1
Orofacial Dyskinesia (Nervous system disorders) | 1
Nose Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Skin Eruption (Skin and subcutaneous tissue disorders) | 1
Thrombosis Venous Deep (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.